CLINICAL TRIAL: NCT04218058
Title: Ultrasound Guided Closed Reduction Versus Open Reduction of Zygomatic Arch in Zygomaticomaxillary Fractures
Brief Title: Reduction of Zygomatic Arch in Zygomaticomaxillary Fractures
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Tasneem Ahmed Mabrouk Amer, assistant lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0020
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Zygomatic Arch Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (ultrasound guided closed reduction of zygomatic arch)) (Active Comparator): reduction of zygomatic arch guided by ultrasound
  Interventions: Procedure: reduction of zygomatic arch in zygomaticomaxillary complex fracture
- control (open reduction of zygomatic arch) (Active Comparator): open reduction of zygomatic arch through coronal incision
  Interventions: Procedure: reduction of zygomatic arch in zygomaticomaxillary complex fracture

INTERVENTIONS:
Procedure: reduction of zygomatic arch in zygomaticomaxillary complex fracture — ultrasound guided reduction of zygomatic arch
  Other Names: open reduction of zygomatic arch in zygomaticomaxillary complex fracture

SUMMARY:
To compare between ultrasound guided closed reduction and open reduction of zygomatic arch in cases of zygomaticomaxillary fracture.

To evaluate the role of intra-operative ultrasound during zygomatic arch reduction.

To compare between esthetic appearance, orbital movement, wound healing, scaring, and postoperative ocular complications in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with ZMC fractures that require reduction and fixation
* Patients between 20 to 50 years old with no gender predilections

Exclusion Criteria:

* Existence of infection at the fracture line
* Chronic systemic diseases such as metabolic bone disease, immunocompromised status

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-11-23 (Actual)

PRIMARY OUTCOMES:
zygomatic arch reduction | immediate post operative CT scan
  to measure the amount of zygomatic arch reduction on postoperative ct scan and compare it with the normal side

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided